CLINICAL TRIAL: NCT04161976
Title: A Study to Assess the Pharmacokinetics, Glucodynamics, Safety, and Tolerability of LY900027 in Patients With Type 1 Diabetes Mellitus on Continuous Subcutaneous Insulin Infusion Therapy
Brief Title: A Study of LY900027 Given by Insulin Pump to Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17489; J2H-MC-IUAA (Other: Eli Lilly and Company); 2019-002318-37 (EudraCT Number)
Record Dates: First submitted 2019-11-12; First posted 2019-11-13 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY900027 (Experimental): LY900027 administered to participants with type 1 diabetes mellitus (T1DM) using continuous subcutaneous insulin infusion (CSII) in one of two dosing periods.
  Interventions: Drug: LY900027
- Insulin Lispro (Active Comparator): Insulin lispro administered to participants with T1DM using CSII in one of two dosing periods.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900027 — LY900027 administered to participants with T1DM using CSII.
  Arms: LY900027
Drug: Insulin Lispro — Insulin lispro administered to participants with T1DM using CSII.
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro

SUMMARY:
The main purpose of this study is to learn more about a new formulation of insulin lispro when given by an insulin pump to participants with type 1 diabetes mellitus. The study will investigate how the body processes the drug and how the drug affects the body. Information about side effects will be collected. The study will last from six to 12 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1DM for at least 1 year
* Fasting C-peptide ≤0.30 nanomoles per liter (nmol/L)
* Bbody mass index between 18.5 and 33.0 kilograms per square meter (kg/m²)
* Participants should have a glycated hemoglobin of ≤9.0% at screening

Exclusion Criteria:

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Pharmacokinetics (PK): Area Under the Insulin Lispro Curve (AUC) 0 to 5 hours after Bolus Administration Prior to a Mixed Meal Tolerance Text (MMTT) | Day 1 through Day 10 in each dosing period
  PK: AUC after Bolus Administration Prior to a MMTT
PK: Maximum Observed Insulin Lispro Concentration (Cmax) | Day 1 through Day 10 in each dosing period
  PK: C PK: Cmax

SECONDARY OUTCOMES:
Pharmacodynamics (PD): Incremental Area Under the Plasma Glucose Curve Above Baseline Between 0-5 hours After Bolus Infusion | Day 1 through Day 10 in each dosing period
  PD: Incremental Area Under the Plasma Glucose Curve Above Baseline Between 0-5 hours After Bolus Infusion
PD: Total Daily Insulin Dose | Day 1 through Day 10 in each dosing period
  PD: Total Daily Insulin Dose
Duration Until Catheter Failure | Day -1 through Day 10 in each dosing period
  Duration Until Catheter Failure

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No